CLINICAL TRIAL: NCT05717179
Title: Ultrasound to Guide Treatment Decisions in Patients With Rheumatoid Arthritis According to a T2T Approach
Acronym: US-RA-T2T
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Italian Society for Rheumatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: US-RA-T2T
Record Dates: First submitted 2022-12-15; First posted 2023-02-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Arthritis, Rheumatoid; Ultrasound; Treat to Target
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional decision strategy (No Intervention): All patients receive a new course of b-ts-DMARDs, with or without concomitant cDMARD. If a CDAI ≤10 is not achieved after 12 weeks, patients are switched to a bDMARD or tsDMARD. The decision on which b/tsDMARD to use at week 12 is at the discretion of the investigator.
- Clinical plus ultrasound-based decision strategy (Experimental): All patients in this group will be evaluated by ultrasound at 44 joints. In case of clinically-verified plus ultrasound verified inflammation, patients will receive a new b-ts-DMARD while continuing or not background csDMARD(s) therapy. If a CDAI ≤10 is not achieved after 12 weeks, patients are again evaluated by ultrasound at 44 joints. In case clinically-verified plus ultrasound-verified inflammation is present, patients are switched to a bDMARD or tsDMARD. The decision on which b/tsDMARD to use is at the discretion of the investigator. In case clinically-verified plus ultrasound-verified inflammation is absent, patients receive step-up pain therapy while background treatment will be continued.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — At baseline and at weeks 12, 24 and 48, patients will undergo an ultrasound examination of 44 joints by one investigator, who is blinded to the strategic arm and all clinical data. The following joints will be assessed: bilateral wrists (distal radio-ulnar joint, radio-carpal, mid-carpal recesses), 1st - 5th MCP, 1st - 5th PIP, elbows, glenohumeral, acromioclavicular, sternoclavicular, knees, ankles and 1st - 5th MTP. At wrists, MCP and PIP joints, palmar and dorsal sites including synovial recess, extensor and flexor tendons will be investigated whereas at feet the dorsal site (plus the lateral aspects of MTP5) including synovial recess and extensor tendons will be evaluated. Further, we will assess the following: at elbows the dorsal and anterior recess, at shoulders the dorsal recess, at knees the suprapatellar as well as the medial and lateral femoro-tibial recess and at ankles the anterior, lateral and medial recess of the tibiotalar joint.
  Arms: Clinical plus ultrasound-based decision strategy

SUMMARY:
Population

Patients with a diagnosis of Rheumatoid Arthritis (RA), moderate or high clinical disease activity (CDAI>10) despite conventional synthetic (cs)DMARD(s) or bs-ts-DMARDs therapy for ≥3 months, and a maximum of 2 swollen joints (out of 44 joints)

Study design

Randomised multicentre, parallel-arm clinical study

Primary objective

Non-inferiority of the experimental arm (i.e. clinical therapy together with ultrasound guided treatment decision) in comparison to the control arm (clinically guided decision) concerning the proportion of patients reaching low disease activity (CDAI ≤10) and a minimal clinical important improvement (MCII: improvement of ≥6 points if starting from moderate disease activity, any case starting from high disease activity and achieving low disease activity) or remission according to ACR/EULAR index-based remission criteria (CDAI ≤2.8/Boolean remission) at week 24.

Intervention

This is a randomised multicentre, national, parallel-arm clinical study. Patients with a diagnosis of RA, moderate or high clinical disease activity (CDAI>10) despite conventional synthetic (cs)DMARD(s) or b-tsDMARDs therapy for ≥3 months, and a maximum of 2 swollen joints (out of 44 joints) will be included and randomized to one of the following two strategic arms:

1. Clinical decision strategy: All patients receive a new course of b-ts-DMARDs, with or without concomitant cDMARD. If a CDAI ≤10 is not achieved after 12 weeks, patients are switched to a bDMARD or tsDMARD. The decision on which b/tsDMARD to use at week 12 is at the discretion of the investigator.
2. Clinical plus ultrasound-based decision strategy. All patients in this group will be evaluated by ultrasound at 44 joints. In case of clinically-verified plus ultrasound verified inflammation, patients will receive a new b-ts-DMARD while continuing or not background csDMARD(s) therapy. If a CDAI ≤10 is not achieved after 12 weeks, patients are again evaluated by ultrasound at 44 joints. In case clinically-verified plus ultrasound-verified inflammation is present, patients are switched to a bDMARD or tsDMARD. The decision on which b/tsDMARD to use is at the discretion of the investigator. In case clinically-verified plus ultrasound-verified inflammation is absent, patients receive step-up pain therapy while background treatment will be continued.

Sample size

158 patients

Time plan

* Total duration of the study: 72 months
* Active phase for each patient: 48 weeks (24 weeks for the interventional treatment strategy and 24 weeks for follow-up visit)
* Recruitment: 60 months

ELIGIBILITY:
Inclusion Criteria:

1. Classification of RA according to the ACR-EULAR 2010 criteria
2. Age of the patients: 18 to 84 years
3. Patients with moderate or high disease activity according to CDAI (>10)
4. Maximum of 2 clinically swollen joints out of a 44-joint count
5. Current stable treatment with a single csDMARD or bDMARD or tsDMARD for at least 3 months
6. No glucocorticoid therapy or stable glucocorticoid dose for at least 4 weeks and at a maximum dose of 5 mg/day prednisone equivalent.
7. No corticosteroid intraarticular injection within 4 weeks
8. Stable or absent dose of NSAIDs for at least 1 week
9. Patients able and willing to give written informed consent and compliant with the requirements of the study protocol

Exclusion Criteria:

1. Complete (clinically evident) destruction of any joint to be investigated by ultrasound as judged by the physician
2. Current RA-related vasculitis or other active systemic (i.e. extraarticular) RA-manifestation except for rheumatoid nodules, which in the opinion of the investigator would expose the study subject to a high risk of morbidity or mortality
3. Initial arthritis manifestations before the age of 18 years
4. Planned surgery within the study period for any of the joints investigated either clinically or by sonography
5. Current severe medical illness requiring hospitalization
6. Active infection or active malignancy at screening <5 years
7. Any contraindication to b/ts DMARDs according to the "Summary of Product Characteristics"
8. Pregnancy or lactation

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of ultrasound-based decision strategy compared to clinically-based strategy. | 24 weeks
  Non-inferiority of the experimental arm (i.e. clinical plus ultrasound-guided treatment decision) in comparison to the control arm (clinically-guided decision) concerning the proportion of patients reaching low disease activity (CDAI ≤10) and a minimal clinical important improvement (MCII: improvement of ≥6 points if starting from moderate disease activity, any case achieving low disease activity who started from high disease activity) [19] or remission according to ACR/EULAR index-based remission criteria (CDAI ≤2.8/Boolean remission) at week 24.

SECONDARY OUTCOMES:
Comparison of the proportion of patients in low disease activity and MCII or remission according to ACR/EULAR index-based remission criteria at week 12 and 48 | 12 and 48 weeks
Comparison of the proportion of patients in remission according to ACR/EULAR index-based remission criteria (CDAI ≤2.8/Boolean remission, respectively) at week 12, 24 and 48 | 12, 24 and 48 weeks
Comparison of the proportion of patients in remission according to DAS-28 (DAS-28 ≤2.6) or SDAI (≤3.3) at week 12, 24 and 48 | 12, 24 and 48 weeks
Comparison of value of tender joints count at weeks 12, 24 and 48 | 12, 24 and 48 weeks
Comparison of value of swollen joints counts at weeks 12, 24 and 48 | 12, 24 and 48 weeks
Comparison of value of VAS (Visual Analogue Scale) pain at weeks 12, 24 and 48 | 12, 24 and 48 weeks
  Range: 0, better outcome - 100, worse outcome
Comparison of value of VAS (Visual Analogue Scale) Patient Global Assessment of Disease Activity at weeks 12, 24 and 48 | 12, 24 and 48 weeks
  Range: 0, better outcome - 100, worse outcome
Comparison of value of VAS (Visual Analogue Scale) Physician Global Assessment of Disease Activity at weeks 12, 24 and 48 | 12, 24 and 48 weeks
  Range: 0, better outcome - 100, worse outcome
Comparison of value of erythrocyte sedimentation rate (ESR) at weeks 12, 24 and 48 | 12, 24 and 48 weeks
Comparison of value of C reactive protein (CRP) at weeks 12, 24 and 48 | 12, 24 and 48 weeks
Comparison of Health assessment questionnaire (HAQ) score at week 24 and 48 | 24 and 48 weeks
  Range: 0, better outcome - 3, worse outcome
Comparison of Rheumatoid Arthritis Impact of Disease (RAID) score at week 24 and 48 | 24 and 48 weeks
  Range: 0, better outcome - 10, worse outcome
Comparison of Fatigue Assessment Scale (FAS) score at week 24 and 48 | 24 and 48 weeks
  Range: 10, better outcome - 50, worse outcome
Comparison of EuroQol-5 dimensions (EQ5D) score at week 24 and 48 | 24 and 48 weeks
Comparison of the trend of VAS (Visual Analogue Scale) pain across all study visits | 48 weeks
  Absolute and relative change of parameter with respect to the baseline and between different visits
Comparison of the trend of VAS (Visual Analogue Scale) Patient Global Assessment of Disease Activity across all study visits | 48 weeks
  Absolute and relative change of parameter with respect to the baseline and between different visits
Comparison of the trend of Health assessment questionnaire (HAQ) score across all study visits | 48 weeks
  Absolute and relative change of score with respect to the baseline and between different visits
Comparison of the trend of Rheumatoid Arthritis Impact of Disease (RAID) score across all study visits | 48 weeks
  Absolute and relative change of score with respect to the baseline and between different visits
Comparison of the trend of Fatigue Assessment Scale (FAS) score across all study visits | 48 weeks
  Absolute and relative change of score with respect to the baseline and between different visits
Comparison of the trend of EuroQol-5 dimensions (EQ5D) score across all study visits | 48 weeks
  Absolute and relative change of score with respect to the baseline and between different visits
Comparison of the differences in the Sharp van der Heijde Score from baseline to week 48 | 48 weeks
  Range: 0, better outcome - 448, worse outcome
Comparison of patients achieving a PD score of ≤1 (44-joint count) at weeks 12, 24 and 48 | 12, 24 and 48 weeks
Comparison of direct medical costs of treatment arms from baseline to week 24 and 48 | 24 and 48 weeks
  Measurement: Incremental cost-effectiveness ratio (ICER)
Analysis regarding predictors of low disease activity or remission at 12, 24 and 48 weeks in patients treated with ≥1bDMARD as compared to those who receive pain therapy | 12, 24 and 48 weeks
  Investigated predictors: baseline erythrocyte sedimentation rate, baseline C reactive protein, baseline ultrasound score (EULAR-OMERACT combined score)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Sanitaria dell'Alto Adige, Bruneck, Bolzano, Italy

IPD SHARING:
Plan to Share IPD: No